CLINICAL TRIAL: NCT03169023
Title: Scale Down: A Randomized, Controlled Weight Management Intervention for Women With Endometrial Cancer
Brief Title: Scale Down for Endometrial Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: ScaleDown (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201701098
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Endometrial Cancer; Cancer of the Endometrium
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: ScaleDown (only first 16 patients) (Experimental): * Baseline quality of life and image surveys
  * Weigh themselves every day on the provided Wi-Fi Scale
  * Personalized feedback with text message comes as soon as participants step on the scale
  * At the 6 month time period, quality of life and body image surveys will be completed and in-office anthropometric assessments will be completed
  * At the end of 6 months, the participants will also receive the "Enhanced Usual Care Packet" which provides printed material from the American Cancer Society Website
  * Only 16 participants were in this arm because ScaleDown went out of business
  * At 12 month follow-up weight will be abstracted from medical record
  Interventions: Behavioral: ScaleDown; Behavioral: Enhanced Usual Care Packets; Other: 12-Item Short Form Health Survey; Other: International Physical Activity Questionnaire short form; Other: Multidimensional Body Self Relations Questionnaire - Appearance Subscales; Other: Cancer-Related Body Image Scale; Other: Patient Health Questionnaire 9-Item Version
- Arm 2: Enhanced Usual Care (Active Comparator): * Baseline quality of life and image surveys
  * Brief in-person counseling session by a research assistant using the Enhanced Usual Care Handouts from the American Cancer Society website which provides guidelines on healthy eating and exercise
  * At the 6 month time period quality of life and body image surveys will be completed and in-office anthropometric assessments will be completed
  * At 12 month follow-up weight will be abstracted from medical record
  Interventions: Behavioral: Enhanced Usual Care Packets; Other: 12-Item Short Form Health Survey; Other: International Physical Activity Questionnaire short form; Other: Multidimensional Body Self Relations Questionnaire - Appearance Subscales; Other: Cancer-Related Body Image Scale; Other: Patient Health Questionnaire 9-Item Version
- Arm 3: iOTA (Experimental): * Baseline quality of life and image surveys
  * Weigh themselves everyday using the provided Balance High Accuracy Digital Body Fat Scale
  * Health coach will meet one-on-one with each participant (in-person or phone) to review health risk assessment and to choose 3 behavior goals related to healthy eating and physical activity at enrollment, 3 months, and 6 months
  * Self-monitoring via SMS text messaging. Weekly check-ins by text providing data about weight and goals
  * At the 6 month time period quality of life and body image surveys will be completed and in-office anthropometric assessments will be completed
  * At the end of 6 months, the participants will also receive the "Enhanced Usual Care Packet" which provides printed material from the American Cancer Society Website
  * At 12 month follow-up weight will be abstracted from medical record
  Interventions: Behavioral: Enhanced Usual Care Packets; Other: 12-Item Short Form Health Survey; Other: International Physical Activity Questionnaire short form; Other: Multidimensional Body Self Relations Questionnaire - Appearance Subscales; Other: Cancer-Related Body Image Scale; Other: Patient Health Questionnaire 9-Item Version; Behavioral: iOTA

INTERVENTIONS:
Behavioral: ScaleDown — -Participants receives behavioral prompts and daily feedback by text messaging with motivational instructions for specific dietary and behavior modifications
  Arms: Arm 1: ScaleDown (only first 16 patients)
Behavioral: Enhanced Usual Care Packets — -From the American Cancer Society Website
Other: 12-Item Short Form Health Survey — -Measures functional health and well-being from the patient's perspective
Other: International Physical Activity Questionnaire short form — -7 item scale that measures a range of physical activity from vigorous to sedentary over the last 7 days
Other: Multidimensional Body Self Relations Questionnaire - Appearance Subscales — -Gold-standard for the assessment of body image attitudes and contains 34 items
Other: Cancer-Related Body Image Scale — -13 item scale adapted from The Breast - impact of Treatment Scale, which assesses survivors' intrusive thoughts and avoidant behaviors with respect to their bodies since cancer treatment
Other: Patient Health Questionnaire 9-Item Version — -Widely used measure that assesses mood, including an item that screens for suicidality
Behavioral: iOTA — -Washington University based intervention
  Arms: Arm 3: iOTA

SUMMARY:
This proposal will pilot a weight management program for patients with endometrial cancer, the cancer most associated with obesity. If successful, this pilot could be expanded to include obese women with other gynecologic cancers (ovarian and cervical) and could be expanded and adapted for use not only upon completion of treatment, but during chemotherapy or radiation. Furthermore, other obstetricians and gynecologists could use this strategy for obese women as a practical cancer prevention strategy for obesity-associated cancers.

ELIGIBILITY:
Inclusion Criteria:

* Female women 18 years of age or older and with biopsy-proven endometrial cancer.
* BMI greater than or equal to 30 kg/m^2.
* Must be able to read and speak English.
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent for Aim 1 study activities in accordance with institutional and federal guidelines.
* Has completed prior surgical management and adjuvant endometrial cancer treatment, if adjuvant treatment is indicated, prior to starting Aim 1.
* Is not receiving concurrent cytotoxic chemotherapy and/or radiation therapy at time of enrollment AND, if randomized, is not anticipated that the participant will need to receive concurrent cytotoxic chemotherapy and/or radiation therapy at any time during the Aim 1 intervention
* Patients with BMI greater than or equal to 30 kg/m^2 who are undergoing hormonal treatment of endometrial cancer.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy of at least one year
* Must have a phone capable of receiving text messages.

Exclusion Criteria:

* Females under the age of 18 years
* BMI less than 30 kg/m^2
* Must not be participating in another formal weight loss program.
* Must not have any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a participant's ability to give informed consent.
* For participants who are randomized in Aim 1:

  * No uncontrolled serious medical or psychiatric condition(s) that would affect the patient's ability to participate in the interventional study, e.g., uncontrolled hypertension, symptomatic cardiac disease, or severe/uncontrolled depression as indicated by a previously completed Patient Health Questionnaire (PHQ-9) score >9 (Kroenke)
  * No diagnoses of any other invasive malignancy other than endometrial cancer or non-melanoma skin cancer which required active treatment currently or within the last 2 years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2019-02-03 (Actual); Study Completion 2019-02-03 (Actual)

PRIMARY OUTCOMES:
Mean weight loss compared between the two arms | Up to 12 months
  -The purpose will be to obtain estimates for the size of an effect achievable by the experimental intervention in order to power and justify a full-scale trial of a weight management program in women with endometrial cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Hagemann, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zamorano AS, Wilson EM, Liu J, Leon A, Kuroki LM, Thaker PH, McCourt CK, Fuh KC, Powell MA, Mutch DG, Evanoff BA, Colditz GA, Hagemann AR. Text-message-based behavioral weight loss for endometrial cancer survivors with obesity: A randomized controlled trial. Gynecol Oncol. 2021 Sep;162(3):770-777. doi: 10.1016/j.ygyno.2021.06.007. Epub 2021 Jun 14. PMID 34140179
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu